CLINICAL TRIAL: NCT00997204
Title: Open Label, Multicenter Study to Evaluate Safety, Local Tolerability, Convenience, and Efficacy of a Self-Administered Subcutaneous Formulation of Icatibant for the Treatment of Acute Attacks of Hereditary Angioedema
Brief Title: EASSI - Evaluation of the Safety of Self-Administration With Icatibant
Acronym: EASSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Jerini AG (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JE049-3101; 2008-000071-25 (EudraCT Number)
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
Keywords: HAE; Type I HAE; Type II HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Icatibant- Naive Treatment Phase (Experimental): Single subcutaneous injection of icatibant, 30 mg
  Interventions: Drug: Icatibant
- icatibant- Self administration Phase (Experimental): Single subcutaneous injection of icatibant, 30 mg
  Interventions: Drug: Icatibant

INTERVENTIONS:
Drug: Icatibant — Single subcutaneous injection of icatibant, 30 mg
  Other Names: Brand name, Firazyr®

SUMMARY:
This study is being conducted to explore the clinical safety, local tolerability, convenience and effectiveness of self-treatment of hereditary angioedema (HAE) attacks with subcutaneous injections of icatibant.

DETAILED DESCRIPTION:
This Phase IIIb study was multi-center and open-label with a single dose level. Subjects with a documented diagnosis of HAE Type I or II were eligible to participate in this trial. Eligible subjects included those who had received treatment for HAE with icatibant in previous clinical trials, or subjects who had been previously treated with the marketed product Firazyr® and subjects who were naïve to icatibant treatment.

All subjects were trained on the method of self-administration at their enrollment visit (Visit 1).For the training sessions, a syringe pre-filled with 3 mL placebo solution was used in place of icatibant. Comprehensive educational material and instructions including pictograms were developed for the subjects to illustrate the method of self-administration and use of the Patient Diary. The training material provided additional information on how to self-diagnose an HAE attack and how to decide on the necessity to treat.In addition, instructions were provided on what to do in case of a laryngeal attack.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study.

1. Males and females 18 years of age at the time of informed consent
2. Documented diagnosis of HAE Type I or II based on ALL of the following criteria:

   * Family and/or medical history
   * Characteristic attack manifestations, recurrent attacks
   * Historical functional C1-INH <50% normal values
3. Women of childbearing potential must use consistently and correctly a highly effective, adequate method of birth control (failure rate less than 1% per year) - sexual abstinence or have a vasectomised partner during the duration of the study. Hormonal contraception can be continued if verified by a physician that it doesn't affect the course of HAE attacks.
4. Mental and physical condition allowing patients to complete baseline assessment, to self-administer icatibant and to follow other study procedures.
5. Ability to provide signed written informed consent after all aspects of the study have been explained and discussed with the patient.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Participation in a clinical trial of another investigational medicinal product within the past month (except a previous icatibant study).
2. Diagnosis of angioedema other than Type I or Type II HAE.
3. Evidence of symptomatic coronary artery disease based on medical history, in particular, unstable angina pectoris or severe coronary heart disease.
4. Congestive heart failure (NYHA Class 3 and 4).
5. Stroke within the past 6 months.
6. Treatment with angiotensin converting enzyme (ACE) inhibitor.
7. Pregnancy and/or breast-feeding.
8. In the opinion of the investigator: mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
9. In the opinion of the investigator: unlikely to comply with the protocol, for example, uncooperative attitude, inability to return for follow-up visits, or unlikely to complete the study for any reason.
10. In the opinion of the investigator: inability to manage study medication or self-administration of an injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-09-25 (Actual); Primary Completion 2011-06-22 (Actual); Study Completion 2011-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (26):
- Hospital Britanico Unidad de Alergia, Buenos Aires, Argentina
- Universitätsklinik für Dermatologie und Venerologie, Graz, Austria
- Odense Universitetshospital-OUH, Odense, I Og Alergicentret, Denmark
- France (5):
  - Centre Hospitalier Universitaire/ Service de Dermatologie, Angers, Angers Cedex 09
  - Hospital Edouaed Herriot, Lyon, Cedex 03
  - Clinique Universitaire de Medicine/ Centre National de reference, Grenoble, Grenoble Cedex 09
  - Hopital Claude Huriex/ Service de medicine interne, Lille, Lille Cedex
  - Hopital Europeen Georges Pompidou Immunologie Clinique, Paris, Paris Cedex 15
- Germany (4):
  - Universitätsmedizin Berlin, Klinik für Dermatologie, Venerologie und Allergologie, Charité, Berlin
  - Universitäts-Hals-Nasen-Ohren-Klinik Essen, Universität Duisburg-Essen, Essen
  - Klinkum der Johann Wolfgang Goethe-Universitat, Frankfurt am Main
  - Hautklinik und Poliklinik, Universitätsmedizin der Johannes Gutenberg-Universität, Mainz
- Israel (3):
  - Bnai-Zion M.C. Clinical Immunology and Allergy Division, Haifa
  - Tel Aviv Sourasky Medical Center - Allergy Unit, Tel Aviv
  - The Chaim Sheba Medical Center, The Allergy and Clinical Immunology Unit, Tel Litwinsky
- Italy (2):
  - Ospedale Luigi Sacco, Milan
  - Universita degli Studi di Napoli 'Federico II', Napoli
- Spain (4):
  - Hospital Universitario Vall de Hebrón / Sección de Alergia, Escola Infermeria, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Servicio de Alergia, Madrid
  - Hospital Universitario La Fe, Servicio de Alergia, Valencia
- Switzerland (2):
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich / Dermatologische Klinik, Zurich
- United Kingdom (3):
  - Southmead Hospital, Department of Immunology, Bristol
  - Barts & The London NHS Trust, Pathology and Pharmacy Building, London
  - Derriford Combined Laboratory, Department of Clinical Immunology & Allergy, Plymouth

REFERENCES:
- [Derived] Aberer W, Maurer M, Reshef A, Longhurst H, Kivity S, Bygum A, Caballero T, Bloom B, Nair N, Malbran A. Open-label, multicenter study of self-administered icatibant for attacks of hereditary angioedema. Allergy. 2014 Mar;69(3):305-14. doi: 10.1111/all.12303. PMID 24438203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened for entry based on their known medical histories (HAE attacks) and previous exposure to a treatment (naïve or not). 151 were enrolled and trained in the self-administration. 47 of these subjects did not have an acute attack of HAE treated with icatibant during this study and were included in the untreated population.
Groups:
- Naive Subjects/ Naive Treatment Phase: Patients who had never received icatibant before this phase, got treatment of Acute HAE Attack with SC icatibant (30 mg)Administered at Site by Health Care Provider.
- Non-Naive Subjects/ Self-administration Phase: Subjects who had received treatment for HAE with icatibant in previous clinical trials or had been previously treated with the marketed product Firazyr®, got Treatment of Acute HAE Attack with SC icatibant (30 mg)Self-Administered.
Period: Naive Treatment Phase
Arm/Group | Naive Subjects/ Naive Treatment Phase | Non-Naive Subjects/ Self-administration Phase
Started | 25 | 79 (Non-naive patients participated in the study but they were not treated in the naive treatment phase)
Completed | 19 | 0
Not Completed | 6 | 79
Period: Self-administration Phase
Arm/Group | Naive Subjects/ Naive Treatment Phase | Non-Naive Subjects/ Self-administration Phase
Started | 19 | 78 (1 subject did not self-administered icatibant but had a HCP to perform. the data were not included.)
Completed | 19 | 77
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-Naive Patients: Patients who previously treated with icatibant in clinical studies or with commercial Firazyr® and got the treatment during the self-administered phase
- Naive Patients: Patients who had never received icatibant and treated in both the Naive treatment phase and the Self-administered phase
- Total: Total of all reporting groups
Arm/Group | Non-Naive Patients | Naive Patients | Total
Number analyzed (Participants) | 79 | 25 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.607 (13.044) | 44.68 (16.53) | 41.58 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 16 | 68
  Male | 27 | 9 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  France | 6 | 0 | 6
  Argentina | 18 | 5 | 23
  Spain | 9 | 2 | 11
  Denmark | 5 | 0 | 5
  Austria | 9 | 5 | 14
  Israel | 15 | 0 | 15
  Germany | 9 | 5 | 14
  Italy | 1 | 1 | 2
  Switzerland | 1 | 1 | 2
  United Kingdom | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events in Self-treatment of Acute HAE Attacks With s.c. Injections of Icatibant
Description: Clinical safety of self-treatment of acute HAE attacks with s.c. injections of icatibant was assessed by calculating the number of AEs occurred during the study. Only those adverse events occurring up to the earlier of 7 days from the start of the naive phase, study discontinuation and start of the self-administration phase are assessed. The Local Tolerability Assessment tool was used. Subjects and Investigators graded erythema/reddening, swelling, burning, pruritus/itching, warm sensation, and skin pain on a 0 to 3 severity scale.
Time Frame: 7 days from the beginning of each phase
Measure: Number; unit: participants
Groups:
- Naive Subjects Administered Icatibant by Health Care Provider: The first HAE attack of naïve subjects enrolled in the study was treated at the study site, where a Health Care Provider administered icatibant to the subject. 3 subjects (of the original 25 enrolled in the naive treatment phase)self-administered icatibant while observed bu HCP, as opposed to having the HCP perform the injection. these data were not included in the naive treatment safety analyses.
- Subjects Who Self-administered Icatibant (Naive): Naive subjects self-administered the study drug at home or other site convenient to the subject, but not at the investigational site, nor under HCP-supervision.
- Subjects Who Self-administered Icatibant (Non-naive): Non-Naive subjects self-administered the study drug at home or other site convenient to the subject, but not at the investigational site, nor under HCP-supervision.
Arm/Group | Naive Subjects Administered Icatibant by Health Care Provider | Subjects Who Self-administered Icatibant (Naive) | Subjects Who Self-administered Icatibant (Non-naive)
Number analyzed (Participants) | 22 | 19 | 78
participants | 11 | 6 | 27

2. Secondary Outcome: Clinical Efficacy of Self-treatment of Acute HAE Attacks With s.c. Injections of Icatibant, Time to Symptom Relief Using VAS Score for a Single Primary Symptom by Patient Cohort
Description: Subjects assessed angioedema attack symptoms using the visual analogue scale (VAS) for skin pain, skin swelling and abdominal pain. The VAS is a continuous scale comprised of a 100 mm in length line, anchored by 2 verbal descriptors, one for each symptom extreme 0 (no pain) and 100 (worst pain). The respondent is asked to place a mark on the VAS line (any where between 0 and 100 mm) at the point that represents their pain intensity. The score is determined by measuring the distance (mm) on the line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Score interpretation is: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). Symptom relief is defined as at least a 50% reduction in a pre-dose VAS score of 30 mm or greater. The time to onset of symptom relief is defined as the first of 3 consecutive assessments at which symptom relief was observed.
Time Frame: 48 hours post-dose
Measure: Median (Inter-Quartile Range); unit: Hours
Groups:
- Naive Subjects Administered Icatibant by Health Care Provider: The first HAE attack of naïve subjects enrolled in the study was treated at the study site, where a Health Care Provider administered icatibant to the subject.
Arm/Group | Naive Subjects Administered Icatibant by Health Care Provider | Subjects Who Self-administered Icatibant (Naive) | Subjects Who Self-administered Icatibant (Non-naive)
Number analyzed (Participants) | 22 | 19 | 78
Hours | 2.0 [1.0 to 4.2] | 3.1 [2.0 to 4.0] | 2.0 [1.0 to 5.3]

ADVERSE EVENTS:
Time Frame: 7 days from the beginning of each phase
Arm/Group | Naive Subjects Administered Icatibant by Health Care Provider | Subjects Who Self-administered Icatibant (Naive) | Subjects Who Self-administered Icatibant (Non-naive)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19 | 0/78
Other Adverse Events (participants affected / at risk) | 7/22 | 6/19 | 21/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naive Subjects Administered Icatibant by Health Care Provider (N=22) | Subjects Who Self-administered Icatibant (Naive) (N=19) | Subjects Who Self-administered Icatibant (Non-naive) (N=78)
Hereditary Angioedema (Congenital, familial and genetic disorders) | 6 | 3 | 19
Headache (Nervous system disorders) | 1 | 1 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Feeling Hot (General disorders) | 0 | 1 | 0
Local Swelling (General disorders) | 0 | 1 | 0
Edema Peripheral (General disorders) | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less